CLINICAL TRIAL: NCT05318664
Title: Effects of Cryotherapy on Upper Limb Balance Test: Randomized Clinical Trial
Brief Title: Effects of Cryotherapy on Upper Limb Balance Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Flávia Carvalho (Other)
Responsible Party: Sponsor-Investigator, Flávia Carvalho, Principal investigator, São Paulo State University
Organization: São Paulo State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EC001
Record Dates: First submitted 2022-03-22; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Functional Status; Muscle Tone
Keywords: shoulder; cryotherapy; balance
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy (Experimental): 20 minutes of cryotherapy on the dominant shoulder with ice bags
  Interventions: Other: Cryotherapy
- Control (No Intervention): 20 minutes of rest

INTERVENTIONS:
Other: Cryotherapy — 20 minutes of cryotherapy on the dominant shoulder with ice bags
  Arms: Cryotherapy

SUMMARY:
The shoulder joint is commonly used and also stricken by high loads and injuries in sports. One technique in emphasis is cryotherapy, a physiotherapeutical intervention characterized by the use of low temperatures for tissue trauma's rehabilitation. Several studies analysed the effects of cryotherapy and brought important results related to pain and strength reduction, also to muscle contraction speed reduction. Although, considering the risk-benefit from de intervention it's pertinent to observe the presence of deleterious effects, especially the ones that impact on motor function. This scenario has been brought by scientists and currently the main gap from this theme resides on the repercussions of the technique application on functional answers

DETAILED DESCRIPTION:
Eighty participants will receive control (rest) and the experimental condition (cryotherapy), with an interval of 48 hours. The intervention group will undergo: i) assessment, ii) 20 minutes of cryotherapy, iii) reassessment, iv) 20 minutes of rest and v) reassessment, while the control group remains at rest for 20 minutes. Assessments will be composed of shoulder function by the upper quarter y balance test, muscle tone by the myoton pro, skin temperature by a thermographic camera, thermic comfort, perception of balance and beliefs in cryotherapy. Data will be described using mean and standard deviation and compared by Mixed ANOVA (time x intervention) with post Bonferroni tests, with significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 28 years old
* healthy
* no musculoskeletal complaints

Exclusion Criteria:

* failure to follow protocol
* complaints of injury or pain during the assessments

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-25 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
modified Upper Quarter Y Balance Test - mUQYBT) | Change from baseline to 20 minutes
  test for measuring upper extremity reach distance while in a closed-chain position
modified Upper Quarter Y Balance Test - mUQYBT) | Change from baseline to 40 minutes
  test for measuring upper extremity reach distance while in a closed-chain position

SECONDARY OUTCOMES:
Skin temperature | Change from baseline to 20 minutes
  thermographic camera FLIR E-8 XT (FLIR Systems, Sweden)
Skin temperature | Change from baseline to 25 minutes
  thermographic camera FLIR E-8 XT (FLIR Systems, Sweden)
Skin temperature | Change from baseline to 30 minutes
  thermographic camera FLIR E-8 XT (FLIR Systems, Sweden)
Skin temperature | Change from baseline to 35 minutes
  thermographic camera FLIR E-8 XT (FLIR Systems, Sweden)
Skin temperature | Change from baseline to 40 minutes
  thermographic camera FLIR E-8 XT (FLIR Systems, Sweden)
Thermic comfort | Change from baseline to 20 minutes
  a 10cm scale ranging from 0 "very comfortable" and 10 "very uncomfortable" will be used
Thermic comfort | Change from baseline to 40 minutes
  a 10cm scale ranging from 0 "very comfortable" and 10 "very uncomfortable" will be used
Balance perception | Change from baseline to 20 minutes
  a likert scale will be used to answer the question " How good was your balance over the test?" 1=nothing, 2=a little, 3=moderate, 4= a lot, 5=extremely
Balance perception | Change from baseline to 40 minutes
  a likert scale will be used to answer the question " How good was your balance over the test?" 1=nothing, 2=a little, 3=moderate, 4= a lot, 5=extremely
Muscle tone | Change from baseline to 20 minutes
  Muscle tone will be measured in hertz by the MyotonPRO wich has a probe that will be placed perpendicular to the skin surface on the muscle belly previously marked with a pen by the evaluator at the Deltoid;
Muscle tone | Change from baseline to 25 minutes
  Muscle tone will be measured in hertz by the MyotonPRO probe will be placed perpendicular to the skin surface on the muscle belly previously marked with a pen by the evaluator at the Deltoid;
Muscle tone | Change from baseline to 30 minutes
  Muscle tone will be measured in hertz by the MyotonPRO probe will be placed perpendicular to the skin surface on the muscle belly previously marked with a pen by the evaluator at the Deltoid;
Muscle tone | Change from baseline to 35 minutes
  Muscle tone will be measured in hertz by the MyotonPRO probe will be placed perpendicular to the skin surface on the muscle belly previously marked with a pen by the evaluator at the Deltoid;
Muscle tone | Change from baseline to 40 minutes
  Muscle tone will be measured in hertz by the MyotonPRO probe will be placed perpendicular to the skin surface on the muscle belly previously marked with a pen by the evaluator at the Deltoid;
Beliefs | Baseline
  The participants will respond yes or no to the questions "Do you believe that cryotherapy is an effect treatment for acute injuries?" and "Do you believe cryotherapy have deleterious effects on muscle function?"

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Pastre, Study Director — São Paulo State University

IPD SHARING:
Plan to Share IPD: No